CLINICAL TRIAL: NCT03985683
Title: Effects of Carbohydrate Loading With Agility Training on Performance in Tennis Players
Brief Title: Nutrition and Agility Training Effect on Performance in Tennis Players
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: REC/00511 Muhammad Hassan
Record Dates: First submitted 2019-06-11; First posted 2019-06-14 (Actual); Last update posted 2020-04-21 (Actual); Status verified 2020-04

CONDITIONS: Sports Physical Therapy
Keywords: Agility training; Carbohydrate loading; Effects on performance

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): In control group athletes will perform T-Test, Illinois agility test, 30 meter run test and Agility Compass drill test, before and after 6 days of intervention.
  Interventions: Other: agility tests
- Experimental (Nutritional Interventional) (Experimental): In experimental group athletes were given 50 % carbohydrate in first 3 days and 70 % in next 3 days respectively. Average carbohydrates required for athletes are 6 to 10 gram per kilogram per day. T-Test, Illinois agility test, 30 meter run test and Agility Compass drill test will use as baseline assessment and after 6 days of intervention.
  Interventions: Dietary Supplement: Nutritional Interventional

INTERVENTIONS:
Other: agility tests — In control group athletes will perform T-Test, Illinois agility test, 30 meter run test and Agility Compass drill test, before and after 6 days of intervention.
  Arms: Control group
Dietary Supplement: Nutritional Interventional — Athletes were given 50 % carbohydrate in first 3 days and 70 % in next 3 days respectively.T-Test, Illinois agility test, 30 meter run test and Agility Compass drill test, before and after 6 days of intervention.
  Arms: Experimental (Nutritional Interventional)

SUMMARY:
The main aim of this study is to determine the effect of carbohydrate loading with combination of agility training in performance of tennis players as previous studies did not show the combining effects of carbohydrate loading and agility training.Total 60 players will be included in this study from which 30 tennis players are in control group and 30 tennis players in experimental group. Baseline Glucose level will be assessed by Gluco-meter before and after intervention of the study each day. In experimental group 50 % carbohydrate will be given in first 3 days and 70 % in next 3 days respectively. Average carbohydrates required for athletes are 6 to 10 gram per kilogram per day. T-Test, Illinois agility test and Agility Compass drill test will use as baseline assessment and after 6 days of intervention and vertical jump height will be assessed through force plates. In control group T-Test will be performed, Illinois agility test and Agility Compass drill test, after 6 days of intervention and vertical jump height will be assessed through force plates.

DETAILED DESCRIPTION:
Tennis is a popular sport with tens of millions of players participating worldwide. This popularity was one factor leading to the reappearance of tennis as a medal sport at the 1988 Summer Olympics in Seoul, South Korea. The volume of play, combined with the physical demands of the sports, can lead to injuries of the musculoskeletal system. Overall, injury incidence and prevalence in tennis has been reported in a number of investigations. The sport creates specific demands on the musculoskeletal system, with acute injuries, such as ankle sprains, being more frequent in the lower extremity while chronic overuse injuries, such as lateral epicondylitis, are more common in the upper extremity in the recreational player and shoulder pain more common in the high-level player.

Tennis tournaments are quite complex due to their variability in terms of exercise duration and the type of effort required. One feature of competitive tennis is that the season is relatively long and that the ranking system pushes players to compete all year long. During a competition, players must sometimes play one or two matches a day on consecutive days. For many reasons the duration and intensity of these matches are highly variable, but it is not uncommon to see matches continue beyond three hours and various studies have shown a drop in high-level tennis performance during extended matches. Under these conditions, optimum recovery methods are needed to maintain a high level of performance over the duration of a match. Among the strategies used, nutrition appears to be an important element to consider.

The majority of studies on the impact of nutritional strategies on tennis performance have been conducted by taking measurements during or at the end of long matches. Some studies have suggested a beneficial effect of carbohydrates during prolonged tennis matches. However, it is increasingly common for competitive athletes to use sports drinks before, during and after matches to help maintain their performance over the duration of a tournament. Different types of commercial beverages, specifically formulated to meet the needs of athletes before, during or after exercise, have been developed and introduced into the market in recent years.

Performance in most sports is determined by the athlete's technical, physiological and psychological characteristics. The physical aspect will be evaluated with a focus on what limits performance, and how training can be conducted to improve performance. Increasing the amount of aerobic high-intensity training, affects physiological adaptations and performance of trained athlete.

Carbohydrate loading regimens is that 2 to 6 days are required for the attainment of supra normal muscle glycogen levels. Because high rates of glycogen re-synthesis are reported during recovery from exercise of near-maximal intensity and that these rates could in theory allow muscle to attain supra normal glycogen levels in less than 24 hours.

Sheppard and Young proposed a definition of agility as "a rapid whole-body movement with change of velocity or direction in response to a stimulus." Agility as the skills and abilities needed to explosively change movement velocities or modes. Agility can therefore be viewed as a context specific ability, with athletes attempting to maximize their sports performance using effective movement as and when required. This allows a full contextualization of movement and allows differentials between sports to be identified, as well as key task differentials between differing playing positions within the same sport.

Previously study in 2014 concluded that there was a significant effect of CHO supplementation on with post-match concentration being higher at the end of the match This double blind, randomized, controlled crossover study was designed to determine the influence of carbohydrate supplementation (0.5 g•kg-1•h-1) on glycaemia, salivary hormones (cortisol and testosterone) concentration, salivary immunoglobulin A (IgA) concentration, and rating of perceived exertion (RPE) during 3 hours of tennis match play in 12 well-trained tennis players. previously study conducted in 2011 and concluded that speed, agility and quickness training program intervention had a positive effect on power performance in young soccer players.

Carbohydrate loading is widely used in various forms. Sports dietitians recommend that early in the week prior to competition athletes maintain a normal moderate-to-high carbohydrate diet as training gradually tapers. previously conducted a study in 2007 and concluded that the use of sprint training as an applicable training method of improving explosive performance of athletes in general.

The main aim of this study is to determine the effect of carbohydrate loading with combination of agility training in performance of tennis players as previous studies did not show the combining effects of carbohydrate loading and agility training.

ELIGIBILITY:
Inclusion Criteria:

* Pakistani tennis players who had experience of 1 year in national tournaments or international tournaments
* Players who don't have history of open or close wound in last 3 months.
* Tennis players with Body Mass Index (BMI) between 18- 24.9.
* Tennis players with random blood glucose level less than 200 mg/dl.
* Athletes age between 15-25 Years.
* Gender: Male.

Exclusion Criteria:

* Players who suffer from any musculoskeletal injury in last 6 months
* Players with any kind of metabolic disorder will be excluded from study.
* Players already taking carbohydrates with their normal diet will be excluded from study.

Ages: 15 Years to 25 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes
Enrollment: 20 (Actual)
Dates: Start 2019-03-02 (Actual); Primary Completion 2019-07-15 (Actual); Study Completion 2019-07-30 (Actual)

PRIMARY OUTCOMES:
T test | 6th day
  In T test players have to run 40 yards and time will be noted in seconds. Rating starts from >11.5 seconds (poor) to <9.5 seconds (excellent).
Illinios agility test | 6th day
  Player have to run about 60 meters and time will be noted in seconds with rating poor >18.8 seconds and excellent <15.9 seconds.
30 meter run test | 6th day
  Player have to run 30 meters in straight line and time will be recorded in seconds
Agility compass drill test | 6th day
  In this test 5 cones are placed in compass design manner and players have to run from cone 1 and finish running at cone 5 and time will be recorded in seconds

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Faheem Afzal, MSSPT, Principal Investigator — Riphah International University
Locations (2):
- Pakistan (2):
  - Riphah International University, Islamabad, Federal, Pakistan
  - Riphah International University, Islamabad, Federal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Amiri-Khorasani M, Sahebozamani M, Tabrizi KG, Yusof AB. Acute effect of different stretching methods on Illinois agility test in soccer players. J Strength Cond Res. 2010 Oct;24(10):2698-704. doi: 10.1519/JSC.0b013e3181bf049c. PMID 20168255
- [Background] Abrams GD, Renstrom PA, Safran MR. Epidemiology of musculoskeletal injury in the tennis player. Br J Sports Med. 2012 Jun;46(7):492-8. doi: 10.1136/bjsports-2012-091164. Epub 2012 May 25. PMID 22554841
- [Background] Haskell WL, Lee IM, Pate RR, Powell KE, Blair SN, Franklin BA, Macera CA, Heath GW, Thompson PD, Bauman A; American College of Sports Medicine; American Heart Association. Physical activity and public health: updated recommendation for adults from the American College of Sports Medicine and the American Heart Association. Circulation. 2007 Aug 28;116(9):1081-93. doi: 10.1161/CIRCULATIONAHA.107.185649. Epub 2007 Aug 1. PMID 17671237
- [Background] Hornery DJ, Farrow D, Mujika I, Young W. Fatigue in tennis: mechanisms of fatigue and effect on performance. Sports Med. 2007;37(3):199-212. doi: 10.2165/00007256-200737030-00002. PMID 17326696
- [Background] Brink-Elfegoun T, Ratel S, Lepretre PM, Metz L, Ennequin G, Dore E, Martin V, Bishop D, Aubineau N, Lescuyer JF, Duclos M, Sirvent P, Peltier SL. Effects of sports drinks on the maintenance of physical performance during 3 tennis matches: a randomized controlled study. J Int Soc Sports Nutr. 2014 Sep 2;11:46. doi: 10.1186/s12970-014-0046-7. eCollection 2014. PMID 25302057
- [Background] Bangsbo J. Performance in sports--With specific emphasis on the effect of intensified training. Scand J Med Sci Sports. 2015 Dec;25 Suppl 4:88-99. doi: 10.1111/sms.12605. PMID 26589122
- [Background] Fairchild TJ, Fletcher S, Steele P, Goodman C, Dawson B, Fournier PA. Rapid carbohydrate loading after a short bout of near maximal-intensity exercise. Med Sci Sports Exerc. 2002 Jun;34(6):980-6. doi: 10.1097/00005768-200206000-00012. PMID 12048325
- [Background] Jeffreys I. A task-based approach to developing context-specific agility. Strength & Conditioning Journal. 2011;33(4):52-9.
- [Background] Gomes RV, Moreira A, Coutts AJ, Capitani CD, Aoki MS. Effect of carbohydrate supplementation on the physiological and perceptual responses to prolonged tennis match play. J Strength Cond Res. 2014 Mar;28(3):735-41. doi: 10.1519/JSC.0b013e3182a1f757. PMID 23860288
- [Background] Jovanovic M, Sporis G, Omrcen D, Fiorentini F. Effects of speed, agility, quickness training method on power performance in elite soccer players. J Strength Cond Res. 2011 May;25(5):1285-92. doi: 10.1519/JSC.0b013e3181d67c65. PMID 21522073
- [Background] Brukner P. Brukner & Khan's clinical sports medicine: McGraw-Hill North Ryde; 2012.
- [Background] Markovic G, Jukic I, Milanovic D, Metikos D. Effects of sprint and plyometric training on muscle function and athletic performance. J Strength Cond Res. 2007 May;21(2):543-9. doi: 10.1519/R-19535.1. PMID 17530960